CLINICAL TRIAL: NCT04425642
Title: Effects of Parenteral Nutrition in Hematopoietic Stem Cell Transplantation: a Randomized Controlled Trial
Brief Title: Effects of Parenteral Nutrition in HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Deputy Director for research, Raisa Gorbacheva Memorial Research Institute for Pediatric Oncology, Hematology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hsct/pn
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Hematologic Malignancy
Keywords: HSCT; Parenteral nutrition
MeSH Terms: conditions — Hematologic Neoplasms; Hyperphagia | interventions — Glucose; Amino Acids; SMOFlipid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose/Amino acids (Experimental): Patients who will require nutritional support will receive parenteral nutrition consisting of glucose and amino acids according age and weight
  Interventions: Drug: Glucose/Amino acids
- Glucose/Amino acids/Lipids (Experimental): Patients who will require nutritional support will receive parenteral nutrition consisting of glucose, amino acids and lipid emulsions according age and weight
  Interventions: Drug: Glucose/Amino acids/Lipids

INTERVENTIONS:
Drug: Glucose/Amino acids — If indications for parenteral nutrition appear, it's dose will be calculated according patient's age and weight and will consist of glucose and amino acids solutions. To prevent potential complications of parenteral nutrition, the target dose will be reached by the third day of therapy. It will discontinued, when the patient oral food intake will be more than 60% for three consecutive days.
  Other Names: Aminoplasmal E 15% 500mL glass bottle; Aminoplasmal E 10% 500mL glass bottle; Aminoven infant 10% 100mL glass bottle; Nutriflex 48/150 1000mL polyethylene 2-chamber bag; Nutriflex 70/240 1500mL polyethylene 2-chamber bag; Glucose 20% 500mL polyethylene bottle
  Arms: Glucose/Amino acids
Drug: Glucose/Amino acids/Lipids — If indications for parenteral nutrition appear, it's dose will be calculated according patient's age and weight and will consist of glucose, amino acids and lipid emulsions. To prevent potential complications of parenteral nutrition, the target dose will be reached by the third day of therapy. It will discontinued, when the patient oral food intake will be more than 60% for three consecutive days.
  Other Names: Aminoplasmal E 15% 500mL glass bottle; SMOFlipid 20% 100mL, 250mL, 500mL glass bottle; Nutriflex 70/180 lipid 625mL polyethylene 3-chamber bag; Aminoplasmal E 10% 500mL glass bottle; Aminoven infant 10% 100mL glass bottle; Nutriflex 48/150 1000mL polyethylene 2-chamber bag; Nutriflex 70/240 1500mL polyethylene 2-chamber bag; SMOFKabiven 1477mL polyethylene 3-chamber bag; Glucose 20% 500mL polyethylene bottle
  Arms: Glucose/Amino acids/Lipids

SUMMARY:
Nutritional therapy implementation in hematopoietic stem cell transplantation (HSCT) have undergone changes recently due to new conditioning regimen and graft versus disease prophylaxis, novel enteral and parenteral nutrition solutions: the value of enteral nutrition is increasing, the indications for parenteral nutrition are becoming more strict. The study aims to identify the role of parenteral nutrition in the context of rapidly changing supportive care approaches in HSCT

DETAILED DESCRIPTION:
The study is interventional: in children and adolescents (2-17 years), adults with blood malignancy and inherited diseases who underwent autologous or allogeneic HSCT, nutritional status, parenteral nutrition tolerability and effectiveness will be assessed before and one month after HSCT. All patients who require parenteral nutrition will pass randomization via envelope technique - solutions containing glucose/amino acids or glucose/amino acids/lipid emulsions. The results will be compared with a control group which will not receive additional nutritional support. The methods used for measurement of nutritional status are: weight, body mass index, bioimpedance and hand grip strength (for adults only), blood tests, diet amount record.

ELIGIBILITY:
Inclusion Criteria:

* Autologous HSCT
* Allogeneic HSCT
* Patients with indications for parenteral nutrition defined as unable to eat more than 50% of oral food intake due to posttransplant complications which leads to malnutrition and malabsorption
* Signed informed consent
* Age > 2 years

Exclusion Criteria:

- Secondary HSCT

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with low tolerability of different parenteral nutrition schemes in HSCT According CTCAE ver. 5.0 | 60 days
  Gastrointestinal toxicity symptoms (anorexia, vomiting, nausea, mucositis, diarrhea) before, during and after discontinuation of parenteral nutrition

SECONDARY OUTCOMES:
Changes in body weight in HSCT depending on nutritional support approach | 30 days
  Changes in body weight (kg) from baseline to day +30
Changes in body mass index in HSCT depending on nutritional support approach | 30 days
  Changes in body mass index (kg/m^2) from baseline to day +30
Changes in body composition in HSCT depending on nutritional support approach | 30 days
  Changes in body composition via bioimpedance by Tanita bc-418 ma, Japan (total body water (kg), muscle mass (kg), fat (kg)) from baseline to day +30
Changes in resting energy expenditure in HSCT depending on nutritional support approach | 30 days
  Changes in resting energy expenditure (kcal) measured via bioimpedance from baseline to day +30 (device - Tanita bc-418 ma, Japan)
Severity and duration of anorexia, nausea, vomiting prevention | 60 days
  According CTCAE ver. 5.0, amount and duration of patient's oral food intake
Impact of parenteral nutrition on infection episodes after HSCT | 60 days
  To compare the incidence of sepsis between patients with and without parenteral nutrition. The sepsis criterions are: laboratory tests - positive blood culture, enchanced serum level of C-reactive protein (mg/L) and procalcitonin (mcg/L); clinical signs - fever.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kulagin, Professor, Study Director — Pavlov First Saint Petersburg State Medical University
Locations (1):
- Pavlov First Saint-Petersburg State Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No